CLINICAL TRIAL: NCT05997693
Title: One Month Dual Antiplatelet Therapy With Ticagrelor in Coronary Artery Bypass Graft Patients
Brief Title: One-Month DAPT in CABG Patients
Acronym: ODIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-06026202; 2023-506613-22 (EudraCT Number); 488058 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2023-07-26; First posted 2023-08-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Coronary Disease
MeSH Terms: interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ticagrelor 90 mg + Low-Dose Aspirin (Experimental)
  Interventions: Drug: Ticagrelor 90 MG; Drug: Low-dose aspirin
- Low-Dose Aspirin Alone (Active Comparator)
  Interventions: Drug: Low-dose aspirin

INTERVENTIONS:
Drug: Ticagrelor 90 MG — Ticagrelor 90 mg twice daily taken orally for one month
  Arms: Ticagrelor 90 mg + Low-Dose Aspirin
Drug: Low-dose aspirin — 75-150 mg once daily taken orally

SUMMARY:
The purpose of this study is to compare the effect of ticagrelor plus low-dose aspirin versus low-dose aspirin alone in patients with chronic coronary disease undergoing coronary artery bypass grafting.

DETAILED DESCRIPTION:
A multinational, randomized trial to evaluate the effect of one-month of ticagrelor plus low-dose aspirin, versus low-dose aspirin alone, on the incidence of death, myocardial infarction, stroke, repeat revascularization and graft failure in patients with chronic coronary disease undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Elective first-time CABG with use of ≥1 saphenous vein graft;
* Ability to sign informed consent and comply with all study procedures, including follow-up for at least 5 years.

Exclusion Criteria:

* Any indication for dual antiplatelet therapy, including

  * Acute/recent (within 1 year) ACS (NSTE-ACS or STEMI)
  * Recent PCI requiring continuation of dual antiplatelet therapy after CABG
* Current or anticipated use of oral anticoagulation;
* Paroxysmal, persistent or permanent atrial fibrillation;
* Any concomitant cardiac or non-cardiac procedure;
* Planned cardiac or non-cardiac surgery within one year;
* Preoperative end-organ dysfunction (dialysis, moderate to severe liver failure, respiratory failure), cancer or other non-cardiac comorbidity with a life expectancy <5 years;
* Inability to use the saphenous vein;
* Contraindications to the use of aspirin;
* Contraindications to the use of ticagrelor, including

  * Known hypersensitivity to ticagrelor
  * Active pathological bleeding (including, but not limited to gastrointestinal or intracranial bleeding)
  * History of intracranial hemorrhage
  * Concomitant therapy with strong CYP3A4 inhibitors (eg ketoconazole, clarithromycin, nefazodone, ritonavir, atazanavir)
* Inability to undergo coronary computed tomographic angiography (CCTA);
* Participating in another investigational device or drug study;
* Women of childbearing potential
* Any major perioperative complication including, but not limited to, stroke, TIA, MI, CABG-related bleeding (BARC type 4), sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of time to death, stroke, myocardial infarction, repeat revascularization and any graft failure. | 1 year
  This is a composite endpoint to be compared between groups in a hierarchical order using the win ratio method. The following hierarchy is pre-specified:
  1. Time to all-cause mortality
  2. Time to stroke
  3. Time to myocardial infarction
  4. Time to coronary revascularization
  5. Presence of graft failure at 12-month imaging follow-up or on unscheduled imaging prior to 12 month

SECONDARY OUTCOMES:
Hierarchical composite of time to death, stroke, myocardial infarction, Bleeding Academic Research Consortium (BARC) type 3 bleeding, repeat revascularization and any graft failure. | 1 year
  This is a composite endpoint to be compared between groups in a hierarchical order using the win ratio method. The following hierarchy is pre-specified:
  1. Time to all-cause mortality
  2. Time to stroke
  3. Time to myocardial infarction
  4. Time to BARC 3 bleeding
  5. Time to coronary revascularization
  6. Presence of graft failure at 12-month imaging follow-up
Hierarchical composite of time to death, stroke, myocardial infarction, repeat revascularization and 5-year time-averaged disease-specific (Seattle Angina Questionnaire [SAQ]-7) quality of life (QoL) score | 5 years
  This is a composite endpoint to be compared between groups in a hierarchical order using the win ratio method. The following hierarchy is pre-specified:
  1. Time to all-cause mortality
  2. Time to stroke
  3. Time to myocardial infarction
  4. Time to coronary revascularization
  5. 5-year time-averaged disease-specific QOL (SAQ-7) score
Hierarchical composite of time to death, stroke, myocardial infarction, BARC type 3 bleeding, repeat revascularization and 5-year time-averaged SAQ-7 QoL score. | 5 years
  This is a composite endpoint to be compared between groups in a hierarchical order using the win ratio method. The following hierarchy is pre-specified:
  1. Time to all-cause mortality
  2. Time to stroke
  3. Time to myocardial infarction
  4. Time to BARC 3 bleeding
  5. Time to coronary revascularization
  6. 5-year time-averaged disease-specific QOL (SAQ-7) score

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ruel, MD, MPH, Principal Investigator — Ottawa Heart Institute Research Corporation; Mario Gaudino, MD, PhD, MSCE, Principal Investigator — Weill Medical College of Cornell University
Locations (22):
- United States (3):
  - Englewood Hospital, Englewood, New Jersey
  - NewYork-Presbyterian: Queens Hospital, Flushing, New York
  - Weill Cornell Medicine, New York, New York
- Austria (4):
  - Medical University Innsbruck, Innsbruck, Innsbruck
  - Medical University Graz, Graz
  - Johannes Kepler University Linz, Linz
  - Medical University of Vienna, Vienna
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada
- China (4):
  - Ruijin Hospital: Shanghai Jiao Tong University School of Medicine, Shanghai, China
  - Jilin Heart Hospital, Changchun, Jilian
  - Beijing Anzhen Hospital, Beijing
  - Center China Fuwai Hospital, Beijing
- Germany (7):
  - University Hospital of Düsseldorf, Düsseldorf
  - Westdeutsches Herz- und Gefäßzentrum Essen, Universität Duisburg-Essen, Essen
  - Klinik für Herz- und Gefäßchirurgie - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Freiburg im Breisgau
  - University Hospital Giessen, Giessen
  - Jena University Hospital, Jena
  - LMU Klinikum Campus Großhadern, München
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Sahlgrenska University Hospital Sweden, Gothenburg
  - Skåne University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandner S, Redfors B, Angiolillo DJ, Audisio K, Fremes SE, Janssen PWA, Kulik A, Mehran R, Peper J, Ruel M, Saw J, Soletti GJ, Starovoytov A, Ten Berg JM, Willemsen LM, Zhao Q, Zhu Y, Gaudino M. Association of Dual Antiplatelet Therapy With Ticagrelor With Vein Graft Failure After Coronary Artery Bypass Graft Surgery: A Systematic Review and Meta-analysis. JAMA. 2022 Aug 9;328(6):554-562. doi: 10.1001/jama.2022.11966. PMID 35943473
- [Derived] Sandner S, Gaudino M, Redfors B, Angiolillo DJ, Ben-Yehuda O, Bhatt DL, Fremes SE, Lamy A, Marano R, Mehran R, Pocock S, Rao SV, Spertus JA, Weinsaft JW, Wells G, Ruel M. One-month DAPT with ticagrelor and aspirin for patients undergoing coronary artery bypass grafting: rationale and design of the randomised, multicentre, double-blind, placebo-controlled ODIN trial. EuroIntervention. 2024 Mar 4;20(5):e322-e328. doi: 10.4244/EIJ-D-23-00699. PMID 38436365